CLINICAL TRIAL: NCT04651894
Title: Cross Sectional Relation of Digital Vascular Function Measured by EndoPAT® in elderlY Patients to Arterial Stiffness
Brief Title: Relationship Between Digital Vascular Function Measured by EndoPAT® in elderlY Patients and Arterial Stiffness
Acronym: ENDY
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Laure JOLY, Professor, Central Hospital, Nancy, France
Other Study IDs: 2020PI228
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Arterial Disease; Frail Elderly Syndrome; Stiffness, Vascular; Endothelial Degeneration
Keywords: endothelial dysfunction; elderly; arterial stiffness; pulse wave velocity; geroscience; vascular aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: reactive hyperaemia index measurement — reactive hyperaemia index with EndoPAT®
  Pulse wave velocity measurement with Sphygmocor®
  Other Names: pulse wave velocity measurement

SUMMARY:
Due to the aging of populations worldwide, we observe an increase of age-related diseases and loss of autonomy with consequent personal, social, medical and economic implications. The aging population is a target for geriatric medicine, necessitating the development of specific diagnostic and therapeutic approaches in order to estimate cardio vascular risk in these individuals.

It is thought that arterial stiffening and endothelial dysfunction are among the earliest vascular properties altered with the onset of cardiovascular disease. Moreover aging is characterized by progressive fragmentation and break down of the elastic components of the aortic media, which are partially replaced by highly cross-linked collagen leading to stiffening, dilation, and elongation of the aorta . A major underlying mechanism of these modifications is endothelial dysfunction due to high oxidative stress and low-grade inflammation. Reactive hyperemia index (RHI), a key outcome of peripheral arterial tonometry (PAT) has recently become a reliable tool to measure microvascular endothelial function. Some studies have recently demonstrated the interest to measure in elderly patients arterial stiffness parameters in order to prevent loss of autonomy. This cross sectional study aimed at demonstrating the link between arterial stiffness evaluated by pulse wave velocity and endothelial dysfunction evaluated by RHI to implement the tools of cardio vascular risk evaluation in a population of elderly patients referred in a geriatric day hospital.

DETAILED DESCRIPTION:
This study is a cross sectional monocentric retrospective study in a geriatric day hospital population coming for frailty and cardio vascular evaluation : clinical data of 148 patients hospitalized from April 2018 to December 2019 (20 months) of the Measurement of the ARterial-Cardiac AGEing and prevention evaluation of FRailty (MARCAGE.FR) geriatric day hospital of Nancy were retrospectively analyzed. Eligible patients were those who had benefited from an EndoPAT® measurement and arterial stiffness evaluation and aged over 60 years. Exclusion criteria to analyze aortic pulse wave velocity was the presence of atrial fibrillation and for EndoPAT® a poor quality of the signal. 105 among these 148 patients were finally selected as they present EndoPAT® good signal (reviewed by two operators).

All subjects arrived in a fasting state at the geriatric day hospital where anthropometric, frailty evaluation, hemodynamic and transcutaneous measurements of aortic pulse wave velocity (AoPWV) were performed at rest. Some of them had a cerebral Magnetic resonance imaging (MRI) examination. Participants were requested not to smoke or drink tea or coffee for 30 minutes and to sit quietly for 10 minutes at least, before blood pressure and other hemodynamic parameters were measured. Individuals were considered hypertensive if they had systolic blood pressure (SBP) values > 150 mm Hg and/or diastolic blood pressure (DBP) values > 90 mm Hg or if they were previously diagnosed as hypertensive and treated with one or more antihypertensive drug.

ELIGIBILITY:
Inclusion Criteria :

* age over 60 years
* referred to a day hospital check up
* arterial stiffness evaluation
* peripheral Arterial Tonometry Evaluation

Exclusion Criteria:

* atrial fibrillation during examination
* poor quality of the signals

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 105 among these 148 patients were finally selected as they present ENDOPAT good signal
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
endothelial dysfunction | 20 minutes
  RHI measurement

SECONDARY OUTCOMES:
pulse wave velocity | 10 minutes
  PWV measurement
PAT signal QUALITY | 10 minutes
  2 operators

CONTACTS AND LOCATIONS:
Overall Officials: Laure Joly, Professor, Principal Investigator — University of Lorraine
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided